CLINICAL TRIAL: NCT00885716
Title: Shared Decision Making: Ein Kommunikationstraining für Patienten Mit Schizophrenie
Brief Title: A Shared Decision Making Training for Inpatients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: The German-Israeli Foundation for Scientific Research and Development (Other)
Responsible Party: PD Dr. Johannes Hamann, Technische universität München
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GIF2168-1764.1
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2010-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- communication skills training (Experimental): group training in shared decision making.
  Interventions: Behavioral: patient training in shared decision making
- cognitive training (Active Comparator): standard group training of cognitive skills (Konzentrationstraining)
  Interventions: Behavioral: cognitive training

INTERVENTIONS:
Behavioral: patient training in shared decision making
  Arms: communication skills training
Behavioral: cognitive training
  Arms: cognitive training

SUMMARY:
Patients suffering from schizophrenia who attend the communication skills program engage more deeply in therapeutic reasoning and treatment decisions. This results in stronger preferences to participate, greater perceived involvement and better long term adherence compared to patients who do not attend the training.

ELIGIBILITY:
Inclusion Criteria:

* Male and female inpatients with a diagnosis of schizophrenia/schizoaffective disorder according to ICD 10
* between 18 and 60 years of age are eligible for the study
* informed consent
* inpatients

Exclusion Criteria:

* poor German language skills

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Decision Self Efficacy | post intervention

SECONDARY OUTCOMES:
Adherence to medication | 6 months post intervention
Participation preferences | post intervention
Treatment satisfaction | post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Technische Universität München, München, Germany

REFERENCES:
- [Derived] Hamann J, Mendel R, Meier A, Asani F, Pausch E, Leucht S, Kissling W. "How to speak to your psychiatrist": shared decision-making training for inpatients with schizophrenia. Psychiatr Serv. 2011 Oct;62(10):1218-21. doi: 10.1176/ps.62.10.pss6210_1218. PMID 21969650